CLINICAL TRIAL: NCT06521268
Title: Effects of Inspiratory Muscle Training on Lymphedema Volume, Subcutaneous Tissue Thickness, Upper Extremity Functioning, Sleep Quality, and Quality of Life in Upper Extremity Lymphedema Treatment: a Randomized Controlled Study
Brief Title: Effects of Inspiratory Muscle Training on Lymphedema
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Ugur Cavlak, CLINICAL PROFESSOR, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiruniUnivers
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Lymphedema
Keywords: Lymphedema; Inspiratory muscle training; Decongestive treatment; Physical functioning; Sleep quality; Quality of life
MeSH Terms: conditions — Lymphedema; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Inspiratory muscle training
  Interventions: Other: Inspiratory muscle training; Other: Decongestive treatment
- Group 2 (Active Comparator): Controls
  Interventions: Other: Decongestive treatment

INTERVENTIONS:
Other: Inspiratory muscle training — Inspiratory muscle training
  Other Names: Muscle training
  Arms: Group 1
Other: Decongestive treatment — Decongestive treatment

SUMMARY:
The aim of this study is to examine the effect of inspiratory muscle training on lymphedema volume, subcutaneous tissue thickness, upper extremity functionality and sleep quality in the treatment of upper extremity lymphedema. Two groups included 24 patients with lymphedema will be divided into gropus (intervetion and control) and they will compare each other.

DETAILED DESCRIPTION:
All patients will be treated 5 days a week, 4 weeks, with each session lasting 45-60 minutes. While only decongestive treatment will be applied to the control group, inspiratory muscle training will be given to the interventional group in addition to decongestive treatment. Evaluations of the patients will be made before and after of 4-week treatment program.

ELIGIBILITY:
Inclusion Criteria:

Having been diagnosed with lymphedema in the upper extremity at least 6 months ago

* Having stage 2 lymphedema
* Having a 2-8 cm circumference difference between the affected extremity and the healthy extremity at any reference point
* Being between the ages of 18-60
* Voluntarily agreeing to participate in the study
* Not having received any lymphedema treatment in the last 6 months.
* Not having any physical, respiratory, neurological and/or systemic disease that would prevent participation in the treatment program.

Exclusion Criteria:

Having stage 1 and stage 3 lymphedema

* It has been less than 6 months since the diagnosis of lymphedema was made
* Being under 18 years of age and over 60 years of age
* Having a circumference measurement difference of more than 8 cm and less than 2 cm at any reference point between the affected extremity and the healthy extremity
* Lymphedema or elephantiasis with papilloma, hyperkeratosis
* Uncontrolled hypertension, pulmonary edema, presence of serious cardiovascular disease
* Presence of active metastasis
* Acute inflammatory diseases

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Volumetric Measurement | baseline and immediately after the intervention (in the 5th week)
  to measure volume of the upper extremity in milliliter (increased volume compared to the normal upper extremity- increased score means worse outcome)
Measurement of Subcutaneous Tissue Thickness with Ultrasound (US) | baseline and immediately after the intervention (in the 5th week)
  to measure thickness of the tissue (increased thickness compared to the normal upper extremity- increased score means worse outcome)

SECONDARY OUTCOMES:
VISUAL ANALOG SCALE-VAS | baseline and immediately after the intervention (in the 5th week)
  to measure swelling feel, heaviness of edema, and tension of edema (min. score is 0- max.score is10: higher score means worse outcome)
HAND DYNAMOMETER | baseline and immediately after the intervention (in the 5th week)
  to measure hand grip (in Newton- higher score means better score)
Quick Disabilities Of the Arm,Shoulder And Hand (Quick DASH) | baseline and immediately after the intervention (in the 5th week)
  to measure physical functioning of upper extremities (min. scorre is 0-max.score is 100- higher score means worse outcome)
Respiratory Function Test | before and after the intervention (in the 5th week)
  to measure respiratory parameters (FEV1, FVC- higher score means better)
Intraoral pressure measure | before and after the intervention (in the 5th week)
  to measure Intraoral Pressure parameters (MEP and MIP- higher score means better)
Lymphedema Life Impact Scale - LLIS | before and after the intervention (in the 5th week)
  to measure impact of lymphedema on the survivors with lymphedema (min. score is 18 and max. score is 90- higher score means worse outcome)
Lymph-ICF | before and after the intervention (in the 5th week)
  to describe Lymphoedema Functioning, Disability And Health status of the partifcipants (min. score is 0 and max. score is 290- higher score means worse outcome)
Pittsburgh Sleep Quality Index (PSQI) | before and after the intervention (in the 5th week)
  to measure sleep quality (min. score is 0 and max.score is 21 - higher score means worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: UGUR CAVLAK, Prof., Principal Investigator — Biruni University
Locations (1):
- Faculty of Health Sciences in Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hacard F, Machet L, Caille A, Tauveron V, Georgescou G, Rapeneau I, Samimi M, Patat F, Vaillant L. Measurement of skin thickness and skin elasticity to evaluate the effectiveness of intensive decongestive treatment in patients with lymphoedema: a prospective study. Skin Res Technol. 2014 Aug;20(3):274-81. doi: 10.1111/srt.12116. Epub 2013 Nov 27. PMID 24283509